CLINICAL TRIAL: NCT00376480
Title: Delayed Infusion of Ex Vivo Anergized Peripheral Blood Mononuclear Cells Following CD34 Selected Peripheral Blood Stem Cell Transplantation From a Haploidentical Donor for Patients With Acute Leukemia and Myelodysplasia
Brief Title: Laboratory-Treated Lymphocyte Infusion After Haploidentical Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Eva C. Guinan, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-030; P01CA100265 (NIH); P30CA006516 (NIH); MDA-2005-0695; NCT00475384 (obsolete NCT alias)
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts in transformation; adult acute lymphoblastic leukemia in remission; refractory anemia with excess blasts; refractory anemia; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory; Congenital Abnormalities | interventions — Antilymphocyte Serum; fludarabine phosphate; Methylprednisolone; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- administration of adoptive donor lymphocyte infusion (Experimental): administration of donor lymphocytes made using costimulatory blockade ex vivo
  Interventions: Biological: anti-thymocyte globulin; Biological: peripheral blood lymphocyte therapy; Drug: fludarabine phosphate; Drug: methylprednisolone; Drug: thiotepa; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: in vitro-treated peripheral blood stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: peripheral blood lymphocyte therapy
Drug: fludarabine phosphate
Drug: methylprednisolone
Drug: thiotepa
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving total-body irradiation and chemotherapy, such as thiotepa and fludarabine, before a donor stem cell transplant helps stop the growth of cancer or abnormal cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving methylprednisolone and antithymocyte globulin before transplant and peripheral blood cells that have been treated in the laboratory after transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of laboratory-treated peripheral blood cell infusion after donor stem cell transplant in treating patients with hematologic cancers or other diseases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Establish the feasibility of delayed infusion of ex vivo anergized donor peripheral blood mononuclear cells (PBMC) after CD34 (cluster designation 34)-selected megadose haploidentical hematopoietic stem cell transplantation (HSCT) in patients with hematopoietic cancers or other diseases.
* Determine the feasibility of collecting parental allogeneic stimulator cells to induce anergy to the nonshared donor-recipient haplotype in these patients.
* Determine the feasibility of collecting donor PBMC as a source of T cells for ex vivo anergization.
* Determine the number of transplanted individuals who meet the criteria for proceeding to delayed infusion of ex vivo anergized donor PBMC.
* Establish the safety of delayed infusion of ex vivo anergized donor PBMC by establishing the maximum number of donor T cells that can be infused without unacceptable graft-versus-host disease.

Secondary

* Evaluate, in vitro, the induction and specificity of alloantigen hyporesponsiveness in donor PBMC after ex vivo anergization.
* Assess, in vitro, the function of immune cells engrafted in these patients.
* Assess, in vitro, whether alloantigen hyporesponsive donor T cells are present in these patients.
* Develop, preliminarily, in vitro data on the extent of pathogen-specific immunity and its rate of recovery.
* Describe the patterns of opportunistic infections in these patients.

OUTLINE: This is a multicenter, dose-escalation study of ex vivo anergized allogeneic peripheral blood mononuclear cells (PBMC). Patients who are treated on any dose level except dose level 1 are stratified according to age (under 17 [pediatric] vs 17 and over [adult]).

* Myeloablative conditioning regimen: Patients undergo total-body irradiation twice daily on days -11 to -9. Patients also receive thiotepa IV over 4 hours on days -8 and -7, fludarabine phosphate IV over 30 minutes on days -7 to -3, and anti-thymocyte globulin IV over 8 hours and methylprednisolone IV over 15-30 minutes on days -6 to -3.
* Allogeneic peripheral blood stem cell transplantation (PBSCT): Patients undergo CD34-selected PBSCT on day 0.
* Ex vivo anergized allogeneic PBMC infusion: If cells have engrafted and patients are free of active uncontrolled infection and graft-vs-host disease, patients undergo allogeneic or autologous PBMC infusion on day 35 or 42.

Cohorts of 3-8 patients receive escalating doses of ex vivo anergized allogeneic PBMCs until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 5 or 3 of 8 patients experience dose-limiting toxicity.

After completion of study, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute lymphocytic leukemia

    * In ≥ second complete remission (CR), defined as < 5% blasts in bone marrow (BM) and no active extramedullary disease OR in first CR with any of the following high risk features:

      * History of induction failure
      * Philadelphia chromosome positive
      * t(4;11) by cytogenetic analysis
      * Any infant with MLL rearrangements on cytogenetic analysis
    * No relapse with isolated extramedullary disease after completion of prior treatment
  * Acute myeloid leukemia

    * Failed induction therapy after < 3 courses
    * In ≥ second CR, defined as < 5% blasts in BM and no active extramedullary disease OR in first CR with any of the following high-risk features:

      * History of induction failure = 5q- or monosomy 7 cytogenetic findings
  * Any of the following myelodysplastic syndromes:

    * Refractory anemia (RA) with excess blasts (RAEB) with a high International Prognostic Scoring System (IPSS) score or score of intermediate-1(INT-1) or intermediate-2 (INT-2)
    * RAEB in transformation with INT-1, INT-2, or high IPSS score
    * RA with INT-2 score
* Patients must have a healthy, related donor who is at least genotypically HLA-A, B, C, and DR haploidentical to the patient

  * No suitably matched family donor defined by genotypic or phenotypic identity for ≥ 5/6 A, B, or DR loci
  * No immediately available genotypically matched (6/6) unrelated marrow donor
  * No immediately available umbilical cord blood donor with suitable cell dose after a search ≥ 2 months
  * Patients whose medical condition is at high risk of deteriorating or whose disease is at high risk of progression during a donor search are eligible
* Has a parent with a haplotype that is disparate from that of the donor for the haplotype shared by the patient and parent, but not shared by the patient and donor OR patient is able to donate sufficient autologous cells by peripheral blood draw or unstimulated leukapheresis
* No active CNS disease

PATIENT CHARACTERISTICS:

* Room air O_2 saturation > 95% unless the lungs are involved with disease
* No clinical evidence of pulmonary insufficiency unless the lungs are involved with disease
* AST and ALT < 3 times upper limit of normal (ULN)*
* Bilirubin < 2.0 mg/dL*
* Creatinine < 2 times ULN OR creatinine clearance or glomerular filtration rate > 50% of the lower limit of normal
* LVEF > 45% OR shortening fraction > 20%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection, defined as absence of an infectious diagnosis or (in patients who have had a recent positive infectious diagnosis) the resolution of fever, documentation of negative cultures or antigen testing, continuation or completion of a course of appropriate therapy, and presence of stable to resolving clinical symptoms
* No evidence of HIV infection OR known HIV positivity NOTE: *Does not apply if liver is involved with disease

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior stem cell transplantation
* No other concurrent immunosuppressive therapy

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-06 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of making and administering the adoptive T cell product | from conditioning through administration of anergized cells on day 35-42
  ability to collect sufficient cells, make anergized product with good viability, without contamination and infuse per study toxicity of the conditioning regimen, the likelihood of engraftment, and the subsequent percentage of individuals who would be eligible to receive aDLI were determined.
Safety of administering the adoptive T cell product on day 35-42 post haploidentical transplant | the period from aDLI infusion through D100
  rates of graft failure with CD34 selected product, adverse and severe adverse reactions attributable to infusion of anergized donor cells, including fever, hypotension, acute graft vs host disease, organ dysfunction
Alloreactivity engendered by administering the adoptive T cell product | from cell infusion through day 100
  occurrence and severity of acute GVHD

SECONDARY OUTCOMES:
Efficacy in restoring adaptive immunity | from aDLI thorough 1 year
  incidence of viral infection and type of immune reconstitution by phenotype and function of T cells

CONTACTS AND LOCATIONS:
Overall Officials: Eva Guinan, MD, Study Chair — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davies JK, Brennan LL, Wingard JR, Cogle CR, Kapoor N, Shah AJ, Dey BR, Spitzer TR, de Lima M, Cooper LJ, Thall PF, Champlin RE, Nadler LM, Guinan EC. Infusion of Alloanergized Donor Lymphocytes after CD34-selected Haploidentical Myeloablative Hematopoietic Stem Cell Transplantation. Clin Cancer Res. 2018 Sep 1;24(17):4098-4109. doi: 10.1158/1078-0432.CCR-18-0449. Epub 2018 May 16. PMID 29769208